CLINICAL TRIAL: NCT05549167
Title: Efficacy and Safety of Sirolimus in Children and Adolescents With Juvenile Nasopharyngeal Angiofibroma (JNA)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2022--09
Record Dates: First submitted 2022-08-29; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Juvenile Nasopharyngeal Angiofibroma
Keywords: Juvenile nasopharyngeal angiofibroma; JNA; sirolimus
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-randomized interventional study with a historical control group and pilot phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus 0,8 mg/m2, but <2 mg per day, once a day (QD), per os, oral solution, 1mg/ml, 60 ml Optimal individual dosage of sirolimus will be determined under control of concentration in blood serum. Therapeutic concentration - 5-15 ng/ml. Blood samples will be collected until therapeutic concertation will be achieved in 2 consecutive samples, but no more than 4 samples (on the 4th, 7th, 10th, 14th days of admission).

SUMMARY:
Juvenile nasopharyngeal angiofibroma (JNA) is a pathologically benign yet locally aggressive and destructive tumor that develops in the choana and nasopharynx. Historical treatment of JNA has included embolization, surgical resection, and radiation. mTOR signaling way demonstrated to be involved in regulation of growth and angiogenesis of JNA. Sirolimus, as mTOR inhibitor, is a potential target JNA therapy.

The main purpose of the study is to evaluate the efficacy and safety of sirolimus in children and adolescents with primary or recurrent JNA. Efficacy will be estimated based on dynamics of the JNA progression. Historical control group will be used for comparison as standard therapy.

Due to limited experience of sirolimus in JNA in routine practice, study should be conducted in 2 phases: pilot and extended. Decision regarding extended phase will be based on the results of pilot phase.

DETAILED DESCRIPTION:
Juvenile nasopharyngeal angiofibroma (JNA) is a pathologically benign yet locally aggressive and destructive tumor that develops in the choana and nasopharynx. Historical treatment of JNA has included embolization, surgical resection, and radiation. Inhibition of mTOR signaling proved to be an important point in inhibition of JNA growth and vascularization. Sirolimus (rapamun) is an mTOR inhibitor, still data on sirolimus efficacy and safety in JNA is limited to few clinical cases.

The main purpose of the study is to evaluate the efficacy and safety of sirolimus in children and adolescents with primary or recurrent JNA. Historical control will be used for comparison as standard treatment.

Due to limited experience of sirolimus in JNA in routine practice, study should be conducted in 2 phases: pilot and extended.

The duration of the pilot phase is 3 months. Decision regarding conducting of extended phase will be based on the response to treatment in pilot phase. Response to treatment defined as a reduction of the JNA volume or stable volume or an increase in volume < 20% from the initial one.

In the extended period, duration of treatment for patients with primary JNA will be determined by the response to treatment. In case of the response to the therapy, treatment duration will be up to 9 months (3 courses by 3 months each). In case of JNA increase in volume more than 20% from the initial one (control time points 3 and 6 months), sirolimus therapy will be discontinued and surgical intervention to be provided (according to the investigator's decision). After completion of 9 months' treatment period, all patients with primary JNA will receive surgical treatment. The duration of follow up is 3 years In the group of patients with relapse or progression of JNA, therapy will continue up to 3 years or until loss of the response to the therapy (which the earliest).

Optimal individual dosage of sirolimus will be determined under control of concentration in blood serum. Sirolimus therapeutic concentration - 5-15 ng/ml. Blood samples will be collected until therapeutic concertation will be achieved in 2 consecutive samples, but no more than 4 samples (on the 4th, 7th, 10th, 14th days of sirolimus admission).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of JNA.
* Male gender.
* Age 7-18 years.
* Signed informed consent of the parents or the official representative for patients under 14 years of age, the patient and the patient's parents for persons from 14 to 18 years of age.
* Adequate liver and kidney function.
* Patients with primary JNA
* Patients with tumor volume according to MRI >35 ml. Group A1 (Extended phase:) - patients with decrease or stable tumor volume or an increase in tumor volume < 20 %, after 3 months of sirolimus therapy.

Group A2 (Extended phase:)- patients with an increase in tumor volume> 20 % after 3 months of sirolimus therapy or the presence of other indications for surgical treatment, according to the investigator opinion.

Historical control group - patients with diagnosed primary JNA, received treatment in Dmitry Rogachev's Center in the period from January 1, 2013 to April 15, 2022.

* Group B RECCURRENT JNA, Patients with recurrent JNA after primary surgery, who have not previously received sirolimus therapy.
* Historical control group - patients with diagnosed recurrent JNA, received treatment in Dmitry Rogachev' s Center in the period from January 1, 2013 to April 15, 2022.

Exclusion Criteria:

Hypersensitivity to sirolimus or its analogues. The presence of acute or chronic infections, including opportunistic infections.

Hepatic and/or renal insufficiency. The need for concomitant use of inducers (e.g. rifampicin, rifabutin) or inhibitors (e.g. ketoconazole) of the cytochrome CYP3A4 system Previous therapy with sirolimus or other mTOR inhibitors. Indications to palliative therapy, according to investigator's opinion. Participation in other clinical trials.

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with JNA with positive dynamics | 3 months from study enrollment
  The proportion of patients with JNA with positive dynamics (reduction of tumor volume or stabilization of tumor volume or increase in tumor volume < 20% of the initial)

SECONDARY OUTCOMES:
The proportion of patients with JNA with positive dynamics | 6 months from study enrollment
  Primary JNA: The proportion of patients with JNA with positive dynamics (reduction of tumor volume or stabilization of tumor volume or increase in tumor volume < 20% of the initial one
The proportion of patients with JNA with positive dynamics | 9 months from study enrollment
  The proportion of patients with JNA with positive dynamics (reduction of tumor volume or stabilization of tumor volume or increase in tumor volume < 20% of the initial one
proportion of patients with progression after sirolimus therapy initiation | 3, 6, 9 months from study enrollment
  proportion of patients with progression after sirolimus therapy initiation. Progression define as increase of JNA in volume >20% from initial one.
The number and proportion (%) of patients receiving sirolimus without tumor progression in post-surgery catamnesis. | 6, 12, 18, 24, 30, 36 months of post-surgery catamnesis.
Primary JNA: The number of the severe bleeding cases in the post-surgery period | up to 6 days after surgery intervention
  The number of the severe bleeding cases in the post-surgery period in patients receiving sirolimus and in the historical control group.
The blood loss volume in the surgical intervention and postoperative period | up to 6 days after surgery intervention
  The blood loss volume in the surgical intervention and postoperative period in patients receiving sirolimus and in the historical control group
Number and % of patients requiring hem transfusions in the surgical intervention and/or postoperative periods in patients receiving sirolimus and in the historical control group | up to 6 days after surgery intervention
amount of patients required embolization and completeness of embolization in patients receiving sirolimus and in the historical control group. | 1 day of surgery intervention
The proportion of patients (%) with complete and partial removal of JNA in patients treated with sirolimus and in the historical control group. | 1 day of surgery intervention
Recurrent JNA: The number and proportion (%) of patients with tumor progression (tumor growth in the same location) | 6, 9, 15, 21, 27 and 33 months of sirolimus therapy.
Recurrent JNA: The number and proportion (%) of patients with tumor recurrence (tumor growth in new location) treated with sirolimus and in the historical control group | 6, 9, 15, 21, 27 and 33 months of sirolimus therapy.
Recurrent JNA: The number and proportion (%) of patients required surgery intervention or radiotherapy in patients received sirolimus and in the historical control group | 33 months of sirolimus treatment
ALL patients, received sirolimus: progression free survival | up to 36 months of treatment
  ALL patients, received sirolimus: progression free survival ((recurrent JNA) and follow up (primary JNA))
ALL patients, received sirolimus: quality of nasal breath by NOSE questionnaire | For primary JNA: day 7, 14, month 1, 6 , 9 of sirolimus treatment and months 6, 12, 24, 36 of follow up
ALL patients, received sirolimus: quality of nasal breath by NOSE questionnaire | For recurrent JNA - up to 33 months of sirolimus treatment
ALL patients, received sirolimus: safety monitoring frequency and severity of AEs | For recurrent JNA - up to 33 months of sirolimus treatmen

OTHER OUTCOMES:
Optimization of sirolumus dosage regime: Control of sirolimus concentration in blood serum. Therapeutic concentration - 5-15 ng/ml. | Blood samples will be collected until therapeutic concertation will be achieved in 2 consecutive samples, but no more than 4 samples (on the 4th, 7th, 10th, 14th days of admission).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Pediatric Hematology, Oncology and Immunology, Moscow, Russia